CLINICAL TRIAL: NCT01328665
Title: Evaluating an Expressive Writing Intervention About Communicatively-Restricted Organizational Stressors: A Six-Week Randomized, Controlled Trial
Brief Title: Evaluating an Expressive Writing Intervention About Communicatively-Restricted Organizational Stressors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara University (Other)
Responsible Party: Principal Investigator, Justin P. Boren, Assistant Professor, Santa Clara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCUIRB03282011-1
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Stress Disorder
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expressive Writing (Experimental): Affectionate Writing Intervention for 20 minutes per day, 2 times per week, 6 weeks.
  Interventions: Other: Expressive Writing
- No writing (No Intervention): Control Group -- No writing

INTERVENTIONS:
Other: Expressive Writing — Writing intervention for cognitive appraisal of stressor.
  Arms: Expressive Writing

SUMMARY:
This project evaluates the effectiveness of an intervention sought to reduce the physical effects of stress related to those issues that individuals cannot successfully communicate with anyone about. To do this, the investigators will be implementing a writing intervention over the course of the 6-week study. The investigators will be asking all participants to complete questionnaires over the course of the study period. The investigators are also asking participants to provide a small blood sample (from a fingerstick procedure) at two times during the study as well as saliva samples during that same time. The primary research question asks if this intervention procedure is effective. The investigators are evaluating total cholesterol, high sensitivity c-reactive protein, and cortisol.

ELIGIBILITY:
Inclusion Criteria:

* 110 pounds in weight
* Ability to fast for 8 hours prior to laboratory visit
* Staff member at Santa Clara University
* Certain level of inclusionary pretest stress measure

Exclusion Criteria:

* Hepatitis
* Endocrine Disease
* Kidney or Liver Disease
* Cancer (in any form)
* Cushing's disorder
* Rheumatological disorders
* Respiratory Disorders
* Diabetes
* High blood pressure
* Low blood pressure
* Heart or cardiovascular problems
* Chemotherapy
* Current use of alpha or beta blockers, steroids, or hormone replacements
* Pregnant and/or breastfeeding mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Lipids from baseline | Week 1 and Week 6
  Lipid panel includes total cholesterol, High-density lipoproteins, low-density lipoprotein, and triglycerides.
Change in high-sensitivity c-Reactive Protein from baseline | Week 1 and Week 6
Change in Cortisol Awakening Response from Baseline | Week 1 and Week 6
  Measurement of Salivary Cortisol (hydrocortisone, compound-F) as a maximum difference between awakening and 30 minutes after awakening.

SECONDARY OUTCOMES:
Change in Perceived Global Stress over time | Week 1, Week 3, Week 6
  Psychological measure of stress
Change in Organizational Stress over time | Week 1, Week 3, Week 6
  Psychological measure of stress as a function of organizational involvement.
Change in Perception of Communication Restriction of Stressor over time | Week 1, Week 3, Week 6
  Restrictedness of a communicative stressor

CONTACTS AND LOCATIONS:
Overall Officials: Justin P Boren, Ph.D., Principal Investigator — Santa Clara University
Locations (1):
- Santa Clara University, Health Center, Santa Clara, California, United States

REFERENCES:
- [Background] Floyd, K., Boren, J. P., Hannawa, A. F., Hesse, C., McEwan, B., & Veksler, A. E. (2009). Kissing in marital and cohabiting relationships: Effects on blood lipids, stress, and relationship satisfaction. Western Journal of Communication, 73(2), 113 - 133. doi: 10.1080/10570310902856071